CLINICAL TRIAL: NCT06667830
Title: A Comparative Study of Two Different Physical Exercise Programs to Improve Pain, Functional Status, and Physical Performance in Older Adults With Chronic Musculoskeletal Pain: a Randomized Controlled Trial
Brief Title: Effectiveness Study of an Exercise Program for Older Adults With Chronic Musculoskeletal Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Frederico Mesquita Baptista, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT2
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic musculoskeletal pain; Older adults; Exercise program; Physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical exercise (Active Comparator)
  Interventions: Other: Physical exercise program
- Physical exercise + Neural mobilization (Experimental)
  Interventions: Other: Physical exercise program; Other: Neural mobilization techniques

INTERVENTIONS:
Other: Physical exercise program — The physical exercise program will consist of exercises from three different exercise modalities: aerobic training, balance exercises, and isometric exercises.
Other: Neural mobilization techniques — Neural mobilization techniques for the upper and lower quadrants will be actively performed by participants.
  Arms: Physical exercise + Neural mobilization

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a multimodal physical exercise program for older adults (> 60 years) with chronic musculoskeletal pain. The main question it aims to answer is:

What is the impact of the intervention program on participants´ pain intensity (primary outcome), function, physical performance, and somatosensory function (secondary outcomes)? Participants will be assessed at 3 different moments: initial assessment (T0), at the end of the intervention protocol (10 weeks) (T1) and 3 months after the end of the intervention protocol (T2). The intervention protocol will consist of a multimodal exercise program to be carried out over a period of 10 weeks at a frequency of twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 60 years or older
* People with primary or secondary chronic musculoskeletal pain in any body site
* People able to walk independently

Exclusion Criteria:

* Individuals undergoing surgery in the last 3 months
* Patients with a self-reported diagnoses of infection diseases, dementia, tumor/cancer, stroke, uncontrolled diabetes, or at high risk of developing cardiovascular events
* Those with physical limitations that make it impossible for them to carry out the intervention protocols independently (e.g., wheelchair user)
* Patients who are receiving another physical therapy intervention to treat their pain.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Brief Pain Inventory - It assesses pain intensity and functional interference related to pain in the last week. In addition to these two main aspects, it also evaluates the location of the pain, the use of medications and the amount of pain relief in the last week. The instrument has 4 items relating to pain intensity in the last week and 7 items relating to the functional interference of pain with numerical rating scales (from 0 to 10) where higher values indicate greater pain severity. In situations where the participant reports musculoskeletal pain in more than one site, they will be asked to answer the questions considering their main chronic pain.

SECONDARY OUTCOMES:
Temporal characteristics of pain | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  World Health Organization (WHO) Classification - It is a categorical variable with three different possible response categories: (1) Episodic recurrent pain - recurrent pain attacks with pain-free intervals; (2) Continuous pain - pain is always present; (3) Continuous with pain attacks (recurrent pain flare-ups as exacerbations of ongoing underlying pain).
Neuropathic pain components | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  painDETECT questionnaire - The instrument consists of 4 sections related to: (1) pain intensity in the last 4 weeks; (2) the pain pattern; (3) regions of pain; and (4) presence of neuropathic descriptors. The total score is obtained by adding the scores of the last 3 sections and can vary from 1 to 38. Scores ≤ 12 = the neuropathic mechanism is very unlikely to be present (predominance of the nociceptive mechanism); Scores ≥ 19 = there is a high probability of a predominant neuropathic mechanism; Scores > 12 and < 19 = the presence of a mixed component.
Pain Catastrophizing | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Pain Catastrophizing Scale (PCS) - The instrument has 13 items subdivided into three different subscales: helplessness (items 1, 2, 3, 4, 5, and 12); magnification (items 6, 7, and 13); and rumination (items 8, 9, 10, and 11). All subscales are evaluated on a 5-point Likert scale, from 0 (not at all) to 4 (all the time), where higher scores represent a greater level of catastrophizing.
Fear of Movement | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Tampa Scale for Kinesiophobia - The instrument comprises 13 items rated on a 4-point Likert scale, as follows: (1) strongly disagree; (2) somewhat disagree; (3) somewhat agree; (4) strongly agree. The higher the score, the greater the fear perceived during the execution of the movement.
Signs and symptoms of hypersensitivity of the nervous system | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Central Sensitization Inventory (CSI) - It assesses common symptoms and facilitating factors for hypersensitivity of the nervous system in 25 items. The patient scores each response on a scale from 0 (never) to 4 (always). The final score is obtained by summing the scores of the individual items and can range from 0 to 100, where higher scores mean a worse outcome.
Pressure Pain Threshold measured in three different sites (thenar region of the dominant hand; dorsum of foot on dominant side; region of greatest pain) | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Algometer
Q-sense - Cold and Warm Perception Threshold (thenar region of the dominant hand; dorsum of foot on dominant side; region of greatest pain) | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  It will be assessed using a portable quantitative sensory testing device capable of assessing peripheral sensory nerve function using hot and cold thermal sensory thresholds (Q-sense, Medoc).
Q-sense - Heat Pain Threshold (thenar region of the dominant hand; dorsum of foot on dominant side; region of greatest pain) | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  It will be assessed using a portable quantitative sensory testing device capable of assessing peripheral sensory nerve function (Q-sense, Medoc).
Lower Limb Strength | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Five Times Sit to Stand Test
Grip Strength | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Hand-held dynamometer
Balance | T0: baseline assessment; T1: 10 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Functional Reach Test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Sciences (University of Aveiro), Campus Universitário de Santiago, Agra do Crasto, Edifício 30, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No